CLINICAL TRIAL: NCT00920257
Title: A Phase I, Open-Label, Two-Stage Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Oral AKT Inhibitor GSK2141795 in Subjects With Solid Tumors or Lymphomas
Brief Title: A Phase I, Open-Label, First-Time-In-Human Study of the Oral AKT Inhibitor GSK2141795
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112689
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: oncology; breast cancer; AKT inhibitor; first time in human; lymphoma; endometrial cancer; GSK2141795; solid tumors
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Lymphoma; Endometrial Neoplasms | interventions — GSK2141795

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2141795 (Experimental): Oral GSK214179 given daily to patients with cancer. Groups of approximately three patients will receive GSK2141795 at increasing doses until a maximum tolerated dose is identified.
  Interventions: Drug: GSK2141795

INTERVENTIONS:
Drug: GSK2141795 — GSK2141795 is an oral AKT inhibitor.

SUMMARY:
This study is a first time in human, Phase I, open-label, dose-escalation study of the oral AKT inhibitor GSK2141795 in subjects with solid tumors or lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female, 18 years or older.
* Histologically or cytologically confirmed diagnosis of solid tumor malignancy or lymphoma that is not responsive to standard therapies or for which there is no approved or curative therapy. Subjects with malignancies related to human immunodeficiency virus (HIV) or solid organ transplant are excluded.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Able to swallow and retain oral medication.
* Fasting serum glucose <126 mg/dL.
* Male subjects with a female partner of childbearing potential must have had a prior vasectomy or agree to use adequate contraception from the time of the first dose of GSK2141795 until three months after the last dose of GSK2141795.
* A female subject is eligible to participate if she is of non-child bearing potential, or of child-bearing potential and willing to use adequate birth control
* Adequate organ function
* (Part 2 only - endometrial) Histologically or cytologically confirmed diagnosis of relapsed or metastatic endometrial cancer.
* (Part 2 only - endometrial) No more than two prior cytotoxic chemotherapy regimens in the relapsed or metastatic setting. Targeted agents like bevacizumab are not considered cytotoxic chemotherapy for the purposes of this study
* (Part 2 only, breast) Histologically or cytologically confirmed diagnosis of locally advanced or metastatic breast cancer.
* (Part 2 only, breast) No more than three prior cytotoxic chemotherapy regimens in the metastatic setting. Targeted agents like lapatinib, bevacizumab, and trastuzumab are not considered cytotoxic chemotherapy for the purposes of this study

Exclusion Criteria:

* Chemotherapy, radiotherapy, or immunotherapy within 28 days (or 42 days for prior nitrosoureas or mitomycin C) prior to the first dose of GSK2141795. Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity are permitted with approval of a GSK Medical Monitor if dosing of that chemotherapy is terminated at least 14 days prior to the first dose of GSK2141795.
* Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is longer, preceding the first dose of GSK2141795.
* Current use of a prohibited medication or requires any of these medications during treatment with GSK2141795.
* Current use of anticoagulants at therapeutic levels within seven days prior to the first dose of GSK2141795, including warfarin, low molecular weight heparin and direct thrombin inhibitors. Low dose (prophylactic) anticoagulants such as warfarin, low molecular weight heparin, selective Factor Xa inhibitors or direct thrombin inhibitors are permitted provided that subject's PT and PTT meet entry criteria.
* Presence of active gastrointestinal disease or other condition that could affect gastrointestinal absorption (e.g. malabsorption syndrome) or predispose a subject to gastrointestinal ulceration.
* Current use of any anti-platelet agent (e.g. dipyridamole, clopidogrel) other than aspirin (81 mg daily).
* Any major surgery within the last four weeks of screening.
* Unresolved toxicity (except alopecia) greater than or equal to Grade 2 from previous anti-cancer therapy unless agreed to by a GSK Medical Monitor and the investigator, and where a GSK Medical Monitor and the investigator consider that the ongoing toxicity will not introduce additional risk factors and will not interfere with the study procedures.
* Previously diagnosed diabetes mellitus (type 1 or 2).
* Current use of oral corticosteroids, with the exception of inhaled or topical corticosteroids.
* History of an allogeneic stem cell transplant. Subjects with a history of an autologous stem cell transplant are NOT excluded.
* Any serious or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject safety or with obtaining informed consent.
* Symptomatic or untreated CNS metastases or leptomeningeal involvement. Subjects who were previously treated for these conditions, and are asymptomatic without anti-epileptic medications or steroids for at least 2 months are eligible. Subjects with primary brain tumor are excluded.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
* QTc interval greater than or equal to 470 msecs.
* Other clinically significant ECG abnormalities including 2nd degree (type II) or 3rd degree atrioventricular (AV) block.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within the past 6 months.
* Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Pregnant or Lactating females.
* History of HIV infection; history of hepatitis B or C (subject with evidence of cleared hepatitis B are eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-06-16 (Actual); Primary Completion 2013-04-17 (Actual); Study Completion 2013-04-17 (Actual)

PRIMARY OUTCOMES:
To determine the recommended Phase II dose and schedule of GSK214179 using the following information: safety and tolerability, pharmacokinetic (single and repeat dose administration) and pharmacodynamic data | Continune until disease progression or consent withdrawn

SECONDARY OUTCOMES:
• To explore the clinical efficacy of GSK2141795 in subjects with solid tumor malignancies or lymphomas | Continune until disease progression or consent withdrawn
To characterize the metabolite profile of oral GSK2141795 after repeat dose administration in subjects with solid tumor malignancies or lymphoma | Continune until disease progression or consent withdrawn

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (6):
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Aghajanian C, Bell-McGuinn KM, Burris HA 3rd, Siu LL, Stayner LA, Wheler JJ, Hong DS, Kurkjian C, Pant S, Santiago-Walker A, Gauvin JL, Antal JM, Opalinska JB, Morris SR, Infante JR. A phase I, open-label, two-stage study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of the oral AKT inhibitor GSK2141795 in patients with solid tumors. Invest New Drugs. 2018 Dec;36(6):1016-1025. doi: 10.1007/s10637-018-0591-z. Epub 2018 Apr 3. PMID 29611022
- See also: Results for study 112689 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112689?search=study&study_ids=112689#rs